CLINICAL TRIAL: NCT02412436
Title: An Open-Label, Non-Randomized Study of Pharmacokinetic Interactions Among Depot Medroxyprogesterone Acetate (DMPA), Rifampicin (RIF), and Efavirenz (EFV) in Women Co-infected With Human Immunodeficiency Virus (HIV) and Tuberculosis (TB)
Brief Title: PK Study of Rifampicin Interactions With DMPA and Efavirenz in TB
Acronym: PRIDE-HT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5338; UM1AI068636 (NIH)
Record Dates: First submitted 2015-03-17; First posted 2015-04-09 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: HIV-1 Infection; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A: Depot medroxyprogesterone acetate (Experimental): At study entry/week 0, participants received depot medroxyprogesterone acetate (DMPA) 150 mg administered intramuscularly as a single dose and co-administered with rifampicin (RIF) and efavirenz (EFV).
  Interventions: Drug: Depot medroxyprogesterone acetate

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate — Depot medroxyprogesterone acetate intramuscular injection
  Other Names: DMPA

SUMMARY:
This study was done to evaluate the effect of HIV and TB treatment on a commonly used birth control method. It enrolled women who were infected with HIV and TB and were taking efavirenz (EFV; Sustiva®; an anti-HIV medication), rifampicin (RIF; an anti-TB medication), and isoniazid (INH; an anti-TB medication). The purpose of this study was to find out the best frequency to give depot medroxyprogesterone acetate (DMPA; a hormonal birth control method that is given as a shot every 3 months) in these women. This study also tried to find out if a 150 mg injection of DMPA was effective in preventing ovulation, the process by which the ovaries (the ovaries are part of the female reproductive system) release an egg for fertilization, for 12 weeks in women who are taking EFV and RIF. Another purpose of this study was to find out if it is safe to take RIF, EFV and DMPA at the same time.

DETAILED DESCRIPTION:
Globally, women comprise 52% of all people living with human immunodeficiency virus (HIV). Decisions about contraception in a population of women infected with both tuberculosis (TB) and HIV are of paramount importance. In the setting of the treatment of active TB, preventing pregnancy becomes even more important because it allows women to attain a level of health that will support healthy future pregnancies. Treatment options for TB may be limited in pregnancy because of concerns about teratogenicity. Millions of women around the world use depot medroxyprogesterone acetate (DMPA, trade name Depo-Provera) for prevention of pregnancy. DMPA is an intermediate-acting progesterone-only injectable contraceptive with a high efficacy rate. Unfortunately, DMPA's safety and effectiveness among women co-infected with TB and HIV is unknown since the interactions of TB treatment, combination ART (cART), and DMPA have not been well studied. The results of this study are likely to be applicable to women receiving RIF-containing TB treatment who are not being treated concurrently with EFV as well, given that addition of EFV to RIF is unlikely to increase induction of metabolizing enzymes significantly beyond the induction achieved with RIF alone.

The study population included premenopausal women, 18 to 46 years of age, who were co-infected with HIV and TB. To be eligible to enroll in the study, participants must have been on EFV 600 mg once daily plus two or more nucleoside reverse transcriptase inhibitors (NRTIs) for at least 28 days prior to study entry with no plans to change therapy for the 12 weeks of the study. Women must have been on the continuation phase of active TB treatment (with a minimum of 12 weeks remaining) taking RIF 8-12 mg/kg orally and INH 4-6 mg/kg orally on a 5-day or more per week schedule (or as directed by national guidelines for TB treatment). At study entry/week 0, DMPA 150 mg was administered intramuscularly as a single dose.

Study duration was 12 weeks. Visits occurred at weeks 0, 2, 4, 6, 8, 10, and 12. The key evaluations included physical examination, clinical assessments, hematology, chemistry, HIV RNA, pregnancy testing, plasma progesterone levels, and plasma DMPA concentration levels.

The sample size was 46 participants, of which 42 had to be evaluable. Participants who missed two successive visits prior to week 8 and those who did not complete the week 10 and week 12 clinic visits with available DMPA concentrations and progesterone levels were not evaluable and replaced in the sample size. The final number of participants enrolled was 62 participants, with only 42 evaluable.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection.
* Current tuberculosis infection, confirmed or probable diagnosis.
* Currently stable on EFV-based cART for at least 28 days with no intention to change the regimen during the 12-week study period.
* Currently receiving RIF and Isoniazid (INH)-based TB therapy on at least 5 days per week schedule after completion of the intensive phase of TB treatment (minimum of 8 weeks of TB treatment) and expected to be on TB treatment for a minimum of 12 weeks after enrollment. [Does not exclude the use of ethambutol on study.]
* Premenopausal female with presumed normal ovarian function based on normal menstrual history and absence of previous ovarian dysfunction diagnosis.
* Last menstrual period (LMP) ≤35 days prior to study entry.
* Negative serum or urine-HCG pregnancy test within 30 days prior to study entry and negative pregnancy test at entry at any network-approved laboratory that operates in accordance with Good Clinical Practices and participates in appropriate external quality assurance programs.
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or in vitro fertilization) for the duration of the study. Women of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to use an additional reliable method of contraception while in the study. Acceptable forms of contraceptives include:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Non-hormonal IUD
  * Bilateral tubal ligation
  * Male partner vasectomy
* Laboratory values within 30 days prior to study entry:

  * Absolute neutrophil count ≥500 cells/mm^3
  * Platelet count ≥50,000 platelets/mm^3
  * Hemoglobin ≥8.0 g/dL
  * Aspartate transaminase (AST) and alanine aminotransferase (ALT) <5 x upper limit of normal (ULN)
  * Creatinine ≤1.5 x ULN
  * Total bilirubin ≤2.0 x ULN
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Receipt of DMPA or any other injectable contraceptive within 180 days prior to study entry.
* Receipt of other hormonal contraceptives within 30 days prior to study entry.
* Use of any drugs other than RIF and EFV known to: 1) induce CYP3A4 system within 30 days and to 2) inhibit the CYP3A4 system with one week prior to study entry. [Because ethambutol does not induce or inhibit the CYP3A4 system, its use is consistent with the language in the protocol.]
* ≤40 kg in weight.
* Bilateral oophorectomy.
* Less than 30 days postpartum at study entry.
* Hypersensitivity to DMPA, medroxyprogesterone acetate (MPA), or any of the other ingredients in DMPA.
* Any previous breast cancer diagnosis.
* Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to study entry.
* Karnofsky performance score <70 within 14 days prior to study entry.
* Use of any immunosuppressant medication including systemic corticosteroids within 30 days prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* History of deep venous thrombosis or pulmonary emboli.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosie Mngqibisa, MBChB, MPH, Study Chair — Durban Adult HIV CRS; Susan E. Cohn, MD, MPH, Study Chair — Northwestern University; Jennifer Robinson, MD, MPH, Study Chair — Johns Hopkins University
Locations (5):
- Gaborone Prevention/Treatment Trials CRS (12701), Gaborone, Botswana
- Kenya Medical Research Institute/Center for Disease Control (KEMRI/CDC) CRS (31460), Kisumu, Kenya
- South Africa (2):
  - Durban Adult HIV CRS (11201), Durban
  - Univ. of Witwatersrand CRS (11101), Johannesburg
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Derived] Haas DW, Mngqibisa R, Francis J, McIlleron H, Robinson JA, Kendall MA, Baker P, Mawlana S, Badal-Faesen S, Angira F, Omoz-Oarhe A, Samaneka WP, Denti P, Cohn SE; AIDS Clinical Trials Group A5338 Study Team. Pharmacogenetics of interaction between depot medroxyprogesterone acetate and efavirenz, rifampicin, and isoniazid during treatment of HIV and tuberculosis. Pharmacogenet Genomics. 2022 Jan 1;32(1):24-30. doi: 10.1097/FPC.0000000000000448. PMID 34369424
- [Derived] Mngqibisa R, Kendall MA, Dooley K, Wu XS, Firnhaber C, Mcilleron H, Robinson J, Cramer Y, Rosenkranz SL, Roa J, Coughlin K, Mawlana S, Badal-Faesen S, Schnabel D, Omoz-Oarhe A, Samaneka W, Godfrey C, Cohn SE; A5338 Study Team. Pharmacokinetics and Pharmacodynamics of Depot Medroxyprogesterone Acetate in African Women Receiving Treatment for Human Immunodeficiency Virus and Tuberculosis: Potential Concern for Standard Dosing Frequency. Clin Infect Dis. 2020 Jul 27;71(3):517-524. doi: 10.1093/cid/ciz863. PMID 31504342
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at five ACTG Clinical Research Sites in four countries (two sites from South Africa and one site from each of Botswana, Kenya, and Zimbabwe) between November 2015 and March 2017.
Pre-assignment Details: Of the 85 women screened, 62 were deemed eligible and enrolled into this single-arm study.
Period: Overall Study
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Started | 62
Completed | 44
Not Completed | 18
Not completed — Protocol-mandated Discontinuation | 7
Not completed — Lost to Follow-up | 6
Not completed — Unable to get to clinic | 3
Not completed — Death | 1
Not completed — Not Willing to Adhere to Requirements | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [27 to 37]
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 24
  30-39 years | 25
  40-49 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 62
Region of Enrollment [Count of Participants; unit: Participants]
  Botswana | 7
  Zimbabwe | 8
  Kenya | 12
  South Africa | 35
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 20.8 [18.9 to 24.9]
HIV Antiretroviral Therapy [Count of Participants; unit: Participants] — HIV antiretroviral therapy was classified according to the two types of regimens allowed by the protocol.
  Participants
    EFV + two NRTIs | 62
    EFV + more than two NRTIs | 0
HIV RNA [Count of Participants; unit: Participants] — Population: One participant was missing HIV RNA at baseline due to specimen issues.
  Participants
    < 400 copies/mL: number analyzed (Participants) | 61
    < 400 copies/mL | 52
    => 400 copies/mL: number analyzed (Participants) | 61
    => 400 copies/mL | 9
CD4+ Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 407 [209 to 644]
TB Treatment [Count of Participants; unit: Participants] — Participants were expected to be on the continuation phase of TB treatment for the length of study follow-up.
  Participants
    RIF and INH | 52
    RIF, INH, and ethambutol | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With DMPA Concentrations Below 0.1 ng/mL at Week 12
Description: The percent of participants with plasma DMPA concentrations below 0.1 ng/mL was calculated with an exact Clopper-Pearson 95% confidence interval. Suppression of ovulation generally occurs as long as the DMPA level is => 0.1 ng/mL.
Time Frame: Week 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
percentage of participants | 11.9 [4.0 to 25.6]

2. Primary Outcome: Percent of Participants With Progesterone Levels Above 1 ng/mL at Week 12
Description: The percent of participants with plasma progesterone levels above 1 ng/mL was calculated with an exact Clopper-Pearson 95% confidence interval. Ovulation generally occurs when the progesterone level is > 5 ng/mL. If there were participants with plasma progesterone levels > 1 ng/mL, then the percent of participants with plasma progesterone levels > 5 ng/mL would have been calculated by study week.
Time Frame: Week 12
Population: Participants who did not have progesterone concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
percentage of participants | 0.0 [0.0 to 8.4]

3. Secondary Outcome: Percent of Participants With DMPA Concentrations Below 0.1 ng/mL at Weeks 2, 4, 6, 8, and 10
Description: The percents of participants with plasma DMPA concentrations below 0.1 ng/mL at weeks 2, 4, 6, 8, and 10 were calculated with exact Clopper-Pearson 95% confidence intervals. Suppression of ovulation generally occurs as long as the DMPA level is => 0.1 ng/mL.
Time Frame: Weeks 2, 4, 6, 8, and 10
Population: Participants who did not have a DMPA concentration at the analysis week of interest were excluded from each analysis as appropriate. For example, participants missing a DMPA concentration at week 4 were excluded from the week 4 analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
percentage of participants
  Week 2 DMPA < 0.1 ng/mL: number analyzed (Participants) | 40
  Week 2 DMPA < 0.1 ng/mL | 0.0 [0.0 to 8.8]
  Week 4 DMPA < 0.1 ng/mL: number analyzed (Participants) | 40
  Week 4 DMPA < 0.1 ng/mL | 0.0 [0.0 to 8.8]
  Week 6 DMPA < 0.1 ng/mL: number analyzed (Participants) | 41
  Week 6 DMPA < 0.1 ng/mL | 0.0 [0.0 to 8.6]
  Week 8 DMPA < 0.1 ng/mL | 0.0 [0.0 to 8.4]
  Week 10 DMPA < 0.1 ng/mL | 2.4 [0.1 to 12.6]

4. Secondary Outcome: Cumulative Percentage of Participants With DMPA < 0.1 ng/mL
Description: The cumulative percentage of participants having a DMPA concentration less than 0.1 ng/mL at week 12 was calculated using a Kaplan-Meier estimator with an associated standard error. The confidence interval was calculated using a log-log transformation. Suppression of ovulation generally occurs as long as the DMPA level is => 0.1 ng/mL.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: cumulative percentage of participants
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
cumulative percentage of participants | 11.9 [5.1 to 26.3]

5. Secondary Outcome: DMPA AUC
Description: Describe the DMPA plasma area under the curve (AUC) between 0 and 12 weeks, where AUC(0-12wks) was calculated using non-compartmental methods.The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: ng*week/mL
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
ng*week/mL | 7.63 [5.39 to 11.42]

6. Secondary Outcome: DMPA Cmin
Description: Describe the DMPA minimum observed concentration (Cmin) between 0 and 12 weeks. The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
ng/mL | 0.33 [0.21 to 0.49]

7. Secondary Outcome: DMPA Cmax
Description: Describe the DMPA maximum observed concentration (Cmax) between 0 and 12 weeks. The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
ng/mL | 1.04 [0.67 to 1.66]

8. Secondary Outcome: DMPA CL/F
Description: Describe the apparent DMPA clearance (CL/F) between 0 and 12 weeks. The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: L/week
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
L/week | 19681 [13139 to 27845]

9. Secondary Outcome: Percent of Participants Who Experienced a Grade 3 or Higher Sign/Symptom or Laboratory Abnormality
Description: The percent of participants who experienced a grade 3 (severe) or higher sign/symptom or laboratory abnormality were calculated with an exact Clopper-Pearson 95% confidence interval. Events were graded (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death) according to the DAIDS AE Grading Table (V1.0).
Time Frame: Weeks 2, 4, 6, 8, 10, and 12
Population: All enrolled participants were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 62
percentage of participants | 12.9 [5.7 to 23.9]

10. Secondary Outcome: DMPA Half-life
Description: Describe the terminal elimination half-life of DMPA (t½) between 0 and 12 weeks, where t½ was calculated using nonlinear mixed-effects (NLME) modelling. The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
hours | 55 [23 to 83]

11. Secondary Outcome: Time at Which Participant-specific Estimated Elimination Slopes for DMPA Level Cross the Threshold of 0.1 ng/mL
Description: Describe the time at which DMPA levels drop below the threshold of 0.1 ng/mL, based on participant-specific estimated elimination slopes from nonlinear mixed-effects (NLME) models. The Week 0 time point was drawn prior to DMPA injection.
Time Frame: Weeks 0, 2, 4, 6, 8, 10, and 12
Population: Participants who did not have DMPA concentrations at weeks 10 and 12 were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 42
days | 74.2 [70.1 to 77.6]

ADVERSE EVENTS:
Time Frame: Week 0 to either premature study discontinuation or Week 12
Description: The study protocol required reporting of all new diagnoses; all new signs and symptoms Grade 3 (severe) or higher; all new all Grade 3 or higher laboratory values; and all signs, symptoms, and laboratory values that led to a change in treatment, regardless of grade. Events were graded (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death) according to the DAIDS AE Grading Table (V1.0) and reported per the EAE Manual (V2.0). All enrolled participants were included.
Arm/Group | Arm A: Depot Medroxyprogesterone Acetate
All-Cause Mortality (participants affected / at risk) | 1/62
Serious Adverse Events (participants affected / at risk) | 1/62
Other Adverse Events (participants affected / at risk) | 6/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Depot Medroxyprogesterone Acetate (N=62)
Bicytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Depot Medroxyprogesterone Acetate (N=62)
Neutrophil count decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02412436/Prot_ICF_000.pdf
  • Statistical Analysis Plan: Primary Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT02412436/SAP_001.pdf
  • Statistical Analysis Plan: PK Modeling Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT02412436/SAP_002.pdf